CLINICAL TRIAL: NCT05871931
Title: The Effect of Tidal Model Based Psychiatric Nursing Approach Applied to Mothers of Children Diagnosed With Autism Spectrum Disorder on Internalized Stigma and Psychological Well-Being
Brief Title: The Effect of Tidal Model-Based Psychiatric Nursing Approach on Mothers of Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Zahide Gül YAZGI DEMİR, Principal Investigator, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MERSINU-ZYD-01
Record Dates: First submitted 2023-05-09; First posted 2023-05-23 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder
Keywords: autism spectrum disorder; Tidal Model; internalized stigma; psychological well-being; Psychiatric nursing
MeSH Terms: conditions — Autism Spectrum Disorder; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study, researcher (ZGYD) and participant blinding cannot be performed because the mothers participating in the study know which group they belong to. Upon completion of the study, the data will be transferred to a computer environment and an independent statistician will analyse the data without knowing which group is the intervention group and which is the control group, and the findings will be reported.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tidal Model-based Psychiatric Nursing (Experimental): The intervention group will receive an eight-session Tidal Model-based psychiatric nursing approach. The sessions are planned to take place once a week over an 8-week period. All sessions will be conducted face-to-face.
  Interventions: Other: Tidal Model-based psychiatric nursing approach
- No Intervention: Control Group (No Intervention): No intervention will be applied to the mothers in the control group.

INTERVENTIONS:
Other: Tidal Model-based psychiatric nursing approach — The intervention group will receive an eight-session Tidal Model-based psychiatric nursing approach. The sessions will take place once a week over an 8-week period. All sessions will be conducted face-to-face.
  The content of the interview plan, consisting of a total of 8 interviews, is as follows:
  The first interview was 'Meeting and Pretesting', the second interview was 'Creating a Personal Safety Plan, Making a Holistic Assessment', the third interview was 'Recognizing Emotions, Emotion Management and Communication Skills', the fourth interview was 'Coping Skills', and the fifth interview was 'Self Perception', The sixth interview consisted of 'Strengthening Socialisation', the seventh interview consisted of 'Planning for the Future' and the eighth interview consisted of 'Defining the achievements that will accompany him/her in the next voyages of exploration, ending the relationship between the captain and the lifeguard and making a process evaluation'.
  Arms: Tidal Model-based Psychiatric Nursing

SUMMARY:
The goal of this clinical trial is to examine the effect of Tidal Model-based psychiatric nursing approach on internalized stigma and psychological well-being in mothers of children diagnosed with ASD.

DETAILED DESCRIPTION:
The research will be conducted using a mixed research method that combines qualitative and quantitative research methods. The quantitative part of the research will be conducted using a pre-test-post-test randomised controlled experimental research design, while the qualitative part will be conducted using a phenomenological design.

The study will be conducted with 34 mothers (intervention group = 17, control group = 17) who have children diagnosed with ASD. The intervention group will receive an eight-session Tidal Model-based psychiatric nursing approach. The sessions are planned to take place once a week over an 8-week period. All sessions will be conducted face-to-face. The first and eighth sessions are expected to last an average of 45-50 minutes, while the other sessions are expected to last an average of 70-75 minutes. Personal safety plans, holistic evaluation form , and records of one-on-one sessions will be kept for all sessions conducted. No intervention will be applied to the mothers in the control group. Posttests will be administered to mothers in the intervention group after the eighth interview. Data from the control group will be collected simultaneously with the intervention group. Qualitative data were collected with the metaphor question in the personal information form. The mothers were asked to say "My life story with my child with autism spectrum disorder is like ............. Because ................."" sentence was asked to complete.

ELIGIBILITY:
Inclusion Criteria:

* Having a child diagnosed with ASD who is studying at Karaköprü Special Education and Practice School in Şanlıurfa.
* Those who agree to participate in the research
* No previous diagnosis of mental illness
* 18 years of age or older
* Knowing how to read and write
* The mother who does not have problems in terms of hearing, speaking and understanding that will prevent communication in the interviews.

Exclusion Criteria:

* Under 18 years of age
* Those who have problems in hearing, speaking and understanding that will prevent communication in the interviews
* Mother with any previous diagnosis of mental illness
* Having previously undergone similar intervention
* Having a child with multiple disabilities.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 34 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Parents Internalized Stigma of Mental Illness Scale (PISMI) | Basseline and 8 weeks
  The Internalized Stigma of Mental Illnesses Scale (ISMI) was developed by Boyd-Ritsher et al. (2003), and adapted into Turkish by Ersoy and Varan (2007). Then, by Dikeç et al. (2019) based on ISMI, the scale items were adapted to the parents of individuals with mental illness, and Turkish validity reliability was established. The scale consists of 29 items. The scale includes "alienation (item: 1,5,8,16,17,21)", "confirmation of stereotypes (item: 26,10,18,19,23,29)", "perceived discrimination (item: 3.15)". ,22,25,28)", "social withdrawal (item: 4,9,11,12,13,20)", "resistance to stigma (item: 7,14,24,26,27)" It has five subscales. The items in the scale are answered as "strongly disagree" (1 point), "disagree" (2 points), "agree" (3 points), "strongly agree" (4 points). The scale total score ranges from 29 to 116 and there is no scale cutoff score. A high score from the scale indicates that the internalized stigma of the person is more severe in the negative direction.

SECONDARY OUTCOMES:
Psychological Well-Being Scale (PWS) | Basseline and 8 weeks
  The scale was developed by Diener et al. (2009-2010) and adapted into Turkish by Telef (2013). The scale, which consists of eight items in total, has a seven-point Likert structure (1=Strongly disagree, 2=Disagree, 3=Somewhat disagree, 4=Undecided, 5=Disagree a little, 6=Agree, 7=Strongly agree). All items in the scale are expressed positively and the scale has no sub-dimensions. The lowest score obtained from the scale is 8, and the highest score is 56. The total score obtained from the scale is determined by adding the values given to all the items in the scale. A high score from the scale indicates that the person has a high level of psychological well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Zahide Gül YAZGI DEMİR, PhD Candidate, Principal Investigator — Harran University Vocational School of Health Services; Mualla YILMAZ, Professor, Study Director — Mersin University, Faculty of Nursing
Locations (1):
- Karaköprü Special Education Practice I. Level School, Sanliurfa, Karaköprü, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.